CLINICAL TRIAL: NCT03601494
Title: Perineural Platelet Rich Plasma for Pain and Disability Management in Diabetic Peripheral Neuropathy
Brief Title: Perineural Platelet-rich Plasma for Diabetic Neuropathy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00009919
Record Dates: First submitted 2018-07-12; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Neuropathies; Chronic Pain
Keywords: Diabetic Neuropathies; Chronic pain
MeSH Terms: conditions — Diabetic Neuropathies; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): peri-neural platelet rich plasma injection under ultrasound guidance in addition to medical treatment.
  Interventions: Other: perineural injection of platelet-rich plasma; Drug: medical
- Control (Placebo Comparator): medical treatment only
  Interventions: Drug: medical

INTERVENTIONS:
Other: perineural injection of platelet-rich plasma — Sonographic guided injection was done under complete sterile conditions including skin sterilization, ultrasound probe covered with sterile pad, and a sterile gel. The needle was introduced from the lateral side toward midline using the in-plane approach to target the desired nerve, each nerve was injected by a single dose of 1.5 cc of PRP. Free hand one-man technique was used by the physician who simultaneously managed the ultrasound device by holding the syringe with one hand while scanning the nerve by moving the probe with the other hand. With continuous imaging of the tip of the needle, the syringe was put around the nerve and platelet-rich plasma was injected in the peri-neural tissue.
  Arms: Intervention
Drug: medical — vitamin B complex, α lipoic acid, selective serotonin reuptake inhibitor (SSRI)

SUMMARY:
Peripheral neuropathy is very common in diabetes mellitus (DM). Till now there is no available effective therapy for this pathology. Objective: To evaluate the clinical effect of perineural platelet-rich plasma (PRP) injection as a treatment of diabetic peripheral neuropathy (DPN).

DETAILED DESCRIPTION:
Diabetic Peripheral neuropathy (DPN) is a common complication of diabetes mellitus (DM). Among several complications that contribute to reduce patient's quality of life and life expectancy diabetic neuropathy (DN) generalized or focal leads to an impaired life quality.

The clinical symptoms of DPN range from pain and burning sensations, more at rest or at night; to hypoesthesia or paresthesia, and or numbness.

Different types of peripheral neuropathy are observed in diabetes, axonal or demyelination or both can be present, involves myelinated and un-myelinated, large and small fibers. Nerve conduction studies can detect these changes. Till now, there is no effective therapy for the treatment of DPN.

Since 1950 Platelet-rich plasma (PRP) has been used in dermatology and oral maxillofacial surgery, but its role as an effective alternative treatment in many other clinical applications has been increased over the last years.

Platelets contain more than 1100 proteins, include enzymes, enzyme inhibitors, growth factors, immune messengers, and other bioactive compounds which play a role in tissue repair and wound healing.

Autologous platelet-rich plasma found to promote axon regeneration in studies involving animal models. Platelet derived angiogenesis factors are capable of stimulating new capillary growth by inducing migration of endothelial cells. It was suggested that this was the mechanism by which platelet factors influence the process of angiogenesis and revascularization.

ELIGIBILITY:
Inclusion Criteria:

* type II diabetes mellitus
* diabetic peripheral neuropathy
* six months duration of symptoms,

Exclusion Criteria:

* other causes of neuropathy
* patient refusal
* ulcers or amputations
* peripheral vascular diseases
* vertebral spine disease
* connective tissue disease
* platelet dysfunction syndrome
* critical thrombocytopenia
* local infection
* coagulopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
visual analog scale of pain | 6 months
  it will be measured by visual analog scale

SECONDARY OUTCOMES:
Nerve conduction velocity | 6 months
  changes in nerve conduction velocities in meters/ seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No